CLINICAL TRIAL: NCT04058561
Title: Hospital-Based Cluster Stratified Randomization Control Trial: Determination of Best Magnetically Controlled Growing Rods Implementation Strategy Using Distraction Intervals
Brief Title: Hospital-Based Cluster Trial: Magnetically Controlled Growing Rods Using Distraction Intervals
Acronym: MCGR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pediatric Spine Foundation (Other)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSSG0038
Record Dates: First submitted 2019-08-14; First posted 2019-08-15 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Early-Onset Scoliosis Deformity of Spine
Keywords: Spinal deformity, early onset scoliosis

STUDY DESIGN:
Intervention Model Description: Sites will be randomized into two arms of lengthening intervals: 6 weeks (+/- 2 weeks) or 16 weeks (+/- 2 weeks).
Who Masked: Outcomes Assessor
Masking Description: Radiographs will be uploaded by each site to the coordinating team and will not have access to the information on exposure arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- 6 weeks (Experimental): 6-week lengthening interval
  Interventions: Device: MAGEC® Spinal Bracing And Distraction System
- 16 weeks (Active Comparator): 16-week lengthening interval
  Interventions: Device: MAGEC® Spinal Bracing And Distraction System

INTERVENTIONS:
Device: MAGEC® Spinal Bracing And Distraction System — The magnetically controlled growth rod (MCGR) system is a remotely distractible, magnetically controlled growing rod. The remote capabilities allow for less invasive and less time-consuming outpatient distraction visits, which solves many of the problems facing current growing rod technologies. The MCGR system allows for more frequent lengthenings, and the implanted growing rods can be lengthened more often, which allows MCGR to better approximate normal spine growth compared to Traditional Growing Rods.

SUMMARY:
A hospital-based cluster stratified randomization control study will be conducted to investigate spinal growth in Early Onset Scoliosis patients between 5 and 9 years of age. Patients must have a major coronal curve measuring over 50 degrees and be undergoing Magnetically Controlled Growing Rod treatment. We will be studying 6-week lengthening intervals compared to 16-week lengthening intervals on spinal growth within 3 years.

DETAILED DESCRIPTION:
The Magnetically Controlled Growing Rod (MCGR) system consists of growing rods similarly implanted as with traditional approaches, but with subsequent noninvasive distractions. The implanted growing rods are magnetically controlled and adjusted outside the body using an external remote controller (ERC) following initial surgical insertion. No incision or anesthesia are used for rod lengthening procedures and they are performed by the surgeon in an outpatient or office setting. The purpose of this study is to determine the effect of a 6-week lengthening interval compared to a 16-week lengthening interval on spinal growth in Early Onset Scoliosis patients between 5 and 9 years of age with a major coronal curve over 50 degrees undergoing MCGR treatment within 3 years.

ELIGIBILITY:
Inclusion Criteria:

* All patients with diagnosis of Early Onset Scoliosis (scoliosis before age 10)
* Between 5 and 9 years of age (5.0 to 9.9 years)
* Major curve greater than 50 degrees at time of index surgery
* Dual-rod Magnetically Controlled Growing Rod implantation only
* Spine or rib-based constructs
* Pre-operative and intra-operative halo gravity traction is allowed

Exclusion Criteria:

* Patients with previous spine surgery, including other growth friendly techniques
* Patients who cannot abide by the study requirements due to geographical or other similar constraints

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 210 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Spinal growth | 3 years
  T1-S1 growth

SECONDARY OUTCOMES:
Complications | 3 years
  Wound related, implant related, intraoperative complications, pseudoarthrosis, neurologic injury/impairment, pulmonary, pain, non-surgical, other
Curve correction | 3 years
  Change in magnitude of coronal spinal curvature from pre-op to post-op at 3 years
Health related quality of life: questionnaire | 3 years
  Early onset scoliosis 24 item questionnaire; This is a patient reported outcome measure for quality of life, parental/financial burden, and satisfaction (4 main domains). There are 11 sub-domains: General health, pain/discomfort, pulmonary function, transfer, physical function, daily living, fatigue/energy level, emotion, parental impact, financial impact, and satisfaction. Within satisfaction, there is child and parent satisfaction. The raw score for each item is from 1-5. This can be turned into scale scores of 0-100. The higher values represent a better outcome. Average sub-domain scores as well as domain scores can be calculated.
Burden of care | 3 years
  Early onset scoliosis 24 item questionnaire;This is a patient reported outcome measure for quality of life, parental/financial burden, and satisfaction (4 main domains). There are 11 sub-domains: General health, pain/discomfort, pulmonary function, transfer, physical function, daily living, fatigue/energy level, emotion, parental impact, financial impact, and satisfaction. Within satisfaction, there is child and parent satisfaction. The raw score for each item is from 1-5. This can be turned into scale scores of 0-100. The higher values represent a better outcome. Average sub-domain scores as well as domain scores can be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Vitale, MD, Principal Investigator — Columbia University; Kenneth MC Cheung, MD, FRCS, Principal Investigator — The University of Hong Kong
Locations (20):
- United States (17):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Alfred I. DuPont Hospital for Children, Wilmington, Delaware
  - Children's National Health System, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Children's Physican Group Orthopaedics/Children's Healthcare of Atlanta, Atlanta, Georgia
  - Johns Hopkins University, Baltimore, Maryland
  - C.S. Mott Children's Hospital, University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine, St. Louis Children's Hospital, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Shriners Hospitals for Children - Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Campbell Clinic/Le Bonheur Children's Hospital, Memphis, Tennessee
  - Texas Scottish Rite Hospital, Dallas, Texas
- IWK Health Centre, Halifax, Nova Scotia, Canada
- Turku University Hospital, Department of Pediatric Orthopaedic Surgery, Turku, Finland
- The University of Hong Kong, Department of Orthopaedics and Traumatology, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Corona J, Miller DJ, Downs J, Akbarnia BA, Betz RR, Blakemore LC, Campbell RM Jr, Flynn JM, Johnston CE, McCarthy RE, Roye DP Jr, Skaggs DL, Smith JT, Snyder BD, Sponseller PD, Sturm PF, Thompson GH, Yazici M, Vitale MG. Evaluating the extent of clinical uncertainty among treatment options for patients with early-onset scoliosis. J Bone Joint Surg Am. 2013 May 15;95(10):e67. doi: 10.2106/JBJS.K.00805. PMID 23677368
- [Background] Flynn JM, Matsumoto H, Torres F, Ramirez N, Vitale MG. Psychological dysfunction in children who require repetitive surgery for early onset scoliosis. J Pediatr Orthop. 2012 Sep;32(6):594-9. doi: 10.1097/BPO.0b013e31826028ea. PMID 22892621
- [Background] JAMES JI. Idiopathic scoliosis; the prognosis, diagnosis, and operative indications related to curve patterns and the age at onset. J Bone Joint Surg Br. 1954 Feb;36-B(1):36-49. doi: 10.1302/0301-620X.36B1.36. No abstract available. PMID 13130619
- [Background] Pehrsson K, Larsson S, Oden A, Nachemson A. Long-term follow-up of patients with untreated scoliosis. A study of mortality, causes of death, and symptoms. Spine (Phila Pa 1976). 1992 Sep;17(9):1091-6. doi: 10.1097/00007632-199209000-00014. PMID 1411763
- [Background] Smith JT. The use of growth-sparing instrumentation in pediatric spinal deformity. Orthop Clin North Am. 2007 Oct;38(4):547-52, vii. doi: 10.1016/j.ocl.2007.03.009. PMID 17945134
- [Background] Cheung KM, Cheung JP, Samartzis D, Mak KC, Wong YW, Cheung WY, Akbarnia BA, Luk KD. Magnetically controlled growing rods for severe spinal curvature in young children: a prospective case series. Lancet. 2012 May 26;379(9830):1967-74. doi: 10.1016/S0140-6736(12)60112-3. Epub 2012 Apr 19. PMID 22520264
- [Background] Goldberg CJ, Gillic I, Connaughton O, Moore DP, Fogarty EE, Canny GJ, Dowling FE. Respiratory function and cosmesis at maturity in infantile-onset scoliosis. Spine (Phila Pa 1976). 2003 Oct 15;28(20):2397-406. doi: 10.1097/01.BRS.0000085367.24266.CA. PMID 14560091
- [Background] Thompson GH, Akbarnia BA, Campbell RM Jr. Growing rod techniques in early-onset scoliosis. J Pediatr Orthop. 2007 Apr-May;27(3):354-61. doi: 10.1097/BPO.0b013e3180333eea. PMID 17414025
- [Background] Bess S, Akbarnia BA, Thompson GH, Sponseller PD, Shah SA, El Sebaie H, Boachie-Adjei O, Karlin LI, Canale S, Poe-Kochert C, Skaggs DL. Complications of growing-rod treatment for early-onset scoliosis: analysis of one hundred and forty patients. J Bone Joint Surg Am. 2010 Nov 3;92(15):2533-43. doi: 10.2106/JBJS.I.01471. Epub 2010 Oct 1. PMID 20889912
- [Background] Caldas JC, Pais-Ribeiro JL, Carneiro SR. General anesthesia, surgery and hospitalization in children and their effects upon cognitive, academic, emotional and sociobehavioral development - a review. Paediatr Anaesth. 2004 Nov;14(11):910-5. doi: 10.1111/j.1460-9592.2004.01350.x. PMID 15500489
- [Background] Kain ZN, Mayes LC, O'Connor TZ, Cicchetti DV. Preoperative anxiety in children. Predictors and outcomes. Arch Pediatr Adolesc Med. 1996 Dec;150(12):1238-45. doi: 10.1001/archpedi.1996.02170370016002. PMID 8953995
- [Background] Akbarnia BA, Breakwell LM, Marks DS, McCarthy RE, Thompson AG, Canale SK, Kostial PN, Tambe A, Asher MA; Growing Spine Study Group. Dual growing rod technique followed for three to eleven years until final fusion: the effect of frequency of lengthening. Spine (Phila Pa 1976). 2008 Apr 20;33(9):984-90. doi: 10.1097/BRS.0b013e31816c8b4e. PMID 18427320
- [Background] Feinberg N, Matsumoto H, Hung CW, St Hilaire T, Pawelek J, Sawyer JR, Akbarnia BA, Skaggs DL, Roye BD, Roye DP Jr, Vitale MG. Expert Consensus and Equipoise: Planning a Randomized Controlled Trial of Magnetically Controlled Growing Rods. Spine Deform. 2018 May-Jun;6(3):303-307. doi: 10.1016/j.jspd.2017.11.002. PMID 29735141